CLINICAL TRIAL: NCT05889299
Title: A Phase 1b Proof of Concept Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of OMS906 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Study of the Safety and Efficacy of OMS906 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS906-PNH-002
Record Dates: First submitted 2023-05-04; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OMS906 study drug (Experimental): OMS906 study drug repeat-dose 5 mg/kg SC administration at 4-week intervals
  Interventions: Drug: OMS906 study drug

INTERVENTIONS:
Drug: OMS906 study drug — OMS906 study drug dose repeat-dose 5mg/kg SC administration at 4-week intervals

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy in patients with Paroxysmal Nocturnal Hemoglobinuria (PNH).

DETAILED DESCRIPTION:
This is a Phase 1b, proof of concept, open-label, uncontrolled, fixed-dose study. The primary objective is to assess safety and tolerability of OMS906 in patients with PNH. Patients will receive 5 mg/kg OMS906 administered as subcutaneous (SC) injections at 4-week intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of PNH by flow cytometry with PNH clone size of >10% RBCs and/or granulocytes.
2. Male or female adults 18 years and older.
3. Completed informed consent procedures.
4. Patients who are not receiving complement inhibitor treatment or, alternatively, patients currently treated with eculizumab or ravulizumab with an inadequate response to treatment defined as a Hgb <10.5 g/dL. Patients receiving eculizumab or ravulizumab must be on stable doses for at least 6 months.
5. Hemoglobin level <10.5 g/dL at screening and baseline.
6. Lactate dehydrogenase >1.5 upper limit of normal (ULN) for patients not receiving eculizumab or ravulizumab.
7. Female patients of child-bearing potential (CBP) must have a negative serum test at screening and highly sensitive urine pregnancy test prior to each dose of OMS906.
8. Females must use highly effective birth control to prevent pregnancy during the clinical trial and for 20 weeks (140 days) following their last dose of study drug.
9. Males must use highly effective birth control with a female partner to prevent pregnancy during the clinical trial and for 20 weeks (140 days) following their last dose of study drug.
10. Have received vaccination for Neisseria meningitidis. Patients who have not received this vaccination at the time of screening may be vaccinated at any time prior to 2 weeks before the first study drug administration.

Exclusion Criteria:

1. Treatment with any complement pathway inhibitor except eculizumab or ravulizumab within the 6 months prior to screening.
2. For patients not receiving eculizumab or ravulizumab at the time of screening: receipt of eculizumab within 8 weeks prior to screening or receipt of ravulizumab within 24 weeks prior to screening.
3. History of major organ transplant or hematopoietic stem cell/bone marrow transplant.
4. Reticulocyte count <100,000 /µL, transfusion-free platelet count <30,000/µL or absolute neutrophil count <500 cells/µL at screening.
5. Anemia attributable to any other medical condition apart from PNH.
6. Elevation of liver function tests, defined as total bilirubin >2×ULN, direct bilirubin >1.5xULN, and elevated transaminases, alanine aminotransaminase (ALT) or aspartate transaminase (AST), >2×ULN unless due to PNH related hemolysis.
7. History of any severe hypersensitivity reactions to other monoclonal antibodies or excipients included in the OMS906 preparation.
8. Significant active bacterial, fungal, or viral infection within the 2 weeks of OMS906 drug initiation, including COVID-19 infection.
9. History of primary or secondary immunodeficiency or complement deficiency.
10. Have human immunodeficiency virus, hepatitis B or untreated hepatitis C infection.
11. History of splenectomy.
12. History or prior bacterial meningitis or N. meningitidis infection.
13. Patients on immunosuppressive agents such as but not limited to cyclosporine, mycophenolate mofetil (MMF), tacrolimus, cyclophosphamide, or methotrexate less than 8 weeks prior to first treatment with OMS906 unless on a stable regimen for at least 3 months prior to screening.
14. Patients who require recurrent short courses of systemic corticosteroids (i.e., >4 short courses per year of >2 weeks in duration per course).
15. Pregnant, planning to become pregnant, or nursing female patients.
16. Recent surgery requiring general anesthesia within the 2 weeks prior to screening or expected to have surgery requiring general anesthesia during the Treatment Period.
17. History of any clinically significant medical, neurologic, or psychiatric disorder that in the opinion of the investigator would make the patient unsuitable for participation in the study.
18. Treatment with any investigational medicinal product or investigational device within the 30 days (or within 5x its half-life in days, whichever is the longer period) prior to screening or participation in another concurrent clinical trial involving a therapeutic intervention. Participation in observational studies and/or registry studies is permitted.
19. Unable or unwilling to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess overall safety and tolerability of repeat-dose OMS906 5 mg/kg SC administration at 4-week intervals in patients with PNH. | 48 weeks
  Number of participants with treatment-emergent adverse events assessed by CTCAE v5.0 and changes in laboratory measures, ECGs and physical examination.

SECONDARY OUTCOMES:
To assess preliminary efficacy by the effect on hemolysis and anemia measured by hemoglobin (Hgb). | 48 weeks
  To assess preliminary efficacy by the effect on hemolysis and anemia measured by hemoglobin (Hgb).
To assess preliminary efficacy by the effect on hemolysis and anemia measured by Lactate dehydrogenase (LDH). | 48 weeks
  To assess preliminary efficacy by the effect on hemolysis and anemia measured by Lactate dehydrogenase (LDH).
To assess preliminary efficacy by the effect on hemolysis and anemia measured by red blood cell (RBC) transfusion burden. | 48 weeks
  To assess preliminary efficacy by the effect on hemolysis and anemia measured by red blood cell (RBC) transfusion burden.
To assess preliminary efficacy measured by PK, PD, and ADA. | 48 weeks
  Pharmacokinetics (PK) of multiple-dose administration of OMS906. PK parameters including maximum concentration, area under the time-concentration curve, and terminal half-life. Pharmacodynamics (PD) of multiple-dose administration of OMS906. PD parameters including change from baseline in mature complement factor D (FD) and alternative pathway (AP) activation (ex vivo rabbit RBC lysis). Presence of anti-drug antibodies (ADA) in serum will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (1):
- Omeros Investigational Site, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No